CLINICAL TRIAL: NCT00260247
Title: Induction of Drug Metabolism: A Comparative, Pharmacokinetic in Vivo Study of the Effect of Carbamazepine and Oxcarbazepine on CYP3A4.
Brief Title: Induction of Drug Metabolism: In Vivo Comparison of Carbamazepine and Oxcarbazepine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Danish Research Agency (Other); Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AKF-315
Record Dates: First submitted 2005-11-28; First posted 2005-12-01 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2005-03

CONDITIONS: Metabolic Clearance Rate
Keywords: CYP3A4; Induction; Oxcarbazepine; Carbamazepine; Quinidine; Human; In vivo

INTERVENTIONS:
Drug: carbamazepine oxcarbazepine

SUMMARY:
This is a study of the possible effect of two antiepileptic drug on enzymes in the liver that metabolizes a number of drugs. It is a well know fact that carbamazepine induces some of these enzymes and this may reduce the effect of concomitantly administered drugs. Clinical observations suggest that oxcarbazepine does not induce these enzymes to the same degree.

This study directly compares the ability of these two drugs to induce the cytochrome P450 3A4 enzyme, in healthy volunteers using a well defined biomarker reaction of a specific enzyme activity.

It is the hypothesis that oxcarbazepine induces CYP3A4 to a lesser degree than carbamazepine.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 30
* Non smoker
* No signs or symptoms of disease by routine laboratory analysis, ECG and physical examination (general appearance assessment; pulmonal and cardiac stetoscopy; abdominal palpation)
* Informed consent

Exclusion Criteria:

* signs or symptoms of disease by routine laboratory analysis, ECG and physical examination
* mental disease
* participation in another clinical trial involving drugs with 3 months of randomization
* donation of more than 500 mL blood within 3 months of randomization
* intake of more than 21 alcohol equivanlents (one normal strength beer contain one alcohol equivalent)per week

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Formation clearance of 3-hydroxyquinidine

SECONDARY OUTCOMES:
Ratio of metabolite to drug AUC's of 3-OH quinidine to quinidine.

CONTACTS AND LOCATIONS:
Overall Officials: Per Damkier, MD, Ph.D., Principal Investigator — Odense University Hospital
Locations (1):
- University of Southern Denmark, Odense, Denmark